CLINICAL TRIAL: NCT06043375
Title: Effect of Licorice Root Powder on Parameters of Metabolic Syndrome Related to Polycystic Ovary Syndrome
Brief Title: Evaluation of Licorice Root on Metabolic Syndrome in Polycystic Ovary Syndrome Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Sanaullah Iqbal, professor, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: licorice-PCOS
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Metabolic Syndrome; Polycystic Ovary Syndrome
Keywords: Licorice; Metabolic Syndrome; Polycystic Ovary Syndrome; Licorice Root Powder
MeSH Terms: conditions — Metabolic Syndrome; Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allotted to two groups. One group will receive licorice root powder capsules while the other group will not receive any treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Licorice Root Powder Capsule (Experimental): PCOS diagnosed patients in this group will receive licorice root powder capsules, once per day for 12 weeks.
  Interventions: Dietary Supplement: Licorice Root Powder Capsule
- Control Group (No Intervention): PCOS diagnosed patients in this group will not receive licorice root powder capsules or any treatment for 12 weeks.

INTERVENTIONS:
Dietary Supplement: Licorice Root Powder Capsule — Fresh licorice root will be obtained from local market of Lahore. The root will be washed and dried at room temperature. Then it will be converted into powder using grinder. After sieving the ground powder, it will be filled in capsules. One capsule will contain 1000mg of powder. Participants in experimental group will be instructed to consume one capsule per day.
  Arms: Licorice Root Powder Capsule

SUMMARY:
The goal of this study is to learn about the effect of licorice root powder on parameters of metabolic syndrome in those women diagnosed with PCOS with age range of 15-49 years of age. The study aims to answer the following questions:

* Will licorice root powder consumption will have an impact on parameters of metabolic syndrome which are HDL levels, triglycerides, fasting blood pressure and blood glucose levels and abdominal obesity related to PCOS.
* Will licorice help in lowering stress scores and improve quality of life.

Females with diagnosed PCOS will be recruited in the study and will be randomly allotted to two groups. One group will be intervention group and second will be control group. Participants in intervention group will be given 1000mg of licorice root powder in form of capsules (1 per day). Control group will not take anything. For both groups, SF-12 health survey, and readings of lipid profile, fasting blood glucose and blood pressure and central obesity will be taken. Researcher will compare readings of both groups at baseline and after 3 months of intervention to assess the effect of licorice root powder.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is an endocrine disorder which is characterized by ovarian cyst, irregular menses and elevated androgen levels whereas metabolic syndrome (metS) includes presence of 3 out of 5 conditions which are abdominal obesity, high blood glucose levels, high blood pressure, high triglyceride levels and low HDL levels. Metabolic syndrome and polycystic ovary syndrome have a two-way relationship. The risk of development of metS in PCOS females is five-fold higher than non-PCOS females. If PCOS is not addressed timely then it can lead to infertility. Herbal treatments and ayurvedic medicine is thought to be effective in treating PCOS. A lot of data is available which shows positive results using herbs like cinnamon, aloevera etc but data on licorice root powder is limited. Licorice is one of the oldest herb and has anti-inflammatory, antidiabetic, antiobesity, hypolipidemic and so many other properties which makes it very useful herb.

The objective of this study is to evaluate antidiabetic, hypolipidemic and anti-inflammatory properties of licorice root powder on metabolic syndrome related to PCOS. The study will also observe effect of licorice on stress levels using SF-12 questionnaire.

The study will be conducted in seven steps. Step 1 is the preparation of licorice root powder capsules. Step 2 is recruitment of participants. Participants will be recruited from universities and hospitals after checking their ultrasound report or diagnosis of PCOS by doctor.

Step 3 is dividing the participants into two groups which are control and intervention group based on randomization.

Step 4 is conduction of baseline testing of both groups of abdominal obesity, TGL, HDL, BGL, BP and stress levels.

Step 5 is administration of capsules for 3 months. Step 6 is post-interventional testing. Similar tests will be done as baseline testing.

Step 7 is data analysis. Data will be analyzed using SPSS software and paired sample t test will be used for results interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Females with diagnosed PCOS

Exclusion Criteria:

* Hypertension
* Cardiovascular diseases
* Pregnancy
* Any sort of allergy
* Skin problems
* Females without diagnosed PCOS

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — women of reproductive age (15-49 years)
Enrollment: 55 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Change in abdominal obesity measurement at week 12 | Change from baseline measurement at 3 months
  Abdominal obesity will be assessed using waist circumference measurements. An inches tape will be used to measure waist circumference (normal is less than 80 cm).
Change in fasting blood glucose levels | Change from baseline fasting levels at 3 months
  Fasting blood glucose levels will be measured using glucometer at 8-10 hours of fasting.
Change in fasting blood pressure levels | Change from baseline fasting levels at 3 months
  Fasting blood pressure levels will be measured using sphygmomanometer at 8-10 hours of fasting.
Change in HDL and triglycerides levels | Change from baseline levels at 3 months
  HDL and triglycerides levels will be measured by taking blood sample and running tests in laboratory.

SECONDARY OUTCOMES:
Change in stress levels | Change from baseline test scores at 3 months
  A questionnaire will be used to assess stress levels. SF-12 Health Survey is a validated questionnaire used to assess patients reviews about their health and assessing stress levels using scores. It contains 12 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Sanaullah Iqbal, PhD, Principal Investigator — University of Veterinary and Animal Sciences, Lahore, Punjab, Pakistan.
Locations (1):
- University of Veterinary and Animal Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang H, Ruan X, Li Y, Cheng J, Mueck AO. Oxidative stress indicators in Chinese women with PCOS and correlation with features of metabolic syndrome and dependency on lipid patterns. Arch Gynecol Obstet. 2019 Nov;300(5):1413-1421. doi: 10.1007/s00404-019-05305-7. Epub 2019 Sep 23. PMID 31549221
- [Background] Anjum S, Askari S, Riaz M, Basit A. Clinical Presentation and Frequency of Metabolic Syndrome in Women With Polycystic Ovary Syndrome: An Experience From a Tertiary Care Hospital in Pakistan. Cureus. 2020 Dec 2;12(12):e11860. doi: 10.7759/cureus.11860. PMID 33409094
- [Background] Maffazioli GDN, Lopes CP, Heinrich-Oliveira V, Lobo RA, Hayashida SAY, Soares JM Jr, Maciel GAR, Baracat EC. Prevalence of metabolic disturbances among women with polycystic ovary syndrome in different regions of Brazil. Int J Gynaecol Obstet. 2020 Dec;151(3):383-391. doi: 10.1002/ijgo.13374. Epub 2020 Oct 12. PMID 32931592
- [Background] Shamsi M, Nejati V, Najafi G, Pour SK. Protective effects of licorice extract on ovarian morphology, oocyte maturation, and embryo development in PCOS-induced mice: An experimental study. Int J Reprod Biomed. 2020 Oct 13;18(10):865-876. doi: 10.18502/ijrm.v13i10.7771. eCollection 2020 Oct. PMID 33134799
- [Background] de Medeiros SF, de Medeiros MAS, Barbosa BB, Yamamoto MMW. The Role of Visceral Adiposity Index as Predictor of Metabolic Syndrome in Obese and Nonobese Women with Polycystic Ovary Syndrome. Metab Syndr Relat Disord. 2021 Feb;19(1):18-25. doi: 10.1089/met.2020.0045. Epub 2020 Aug 25. PMID 32845813
- [Background] Zhang Y, Xu Y, Zhang L, Chen Y, Wu T, Liu R, Sui W, Zhu Q, Zhang M. Licorice extract ameliorates hyperglycemia through reshaping gut microbiota structure and inhibiting TLR4/NF-kappaB signaling pathway in type 2 diabetic mice. Food Res Int. 2022 Mar;153:110945. doi: 10.1016/j.foodres.2022.110945. Epub 2022 Jan 10. PMID 35227470
- [Background] Yang JP, Ullah A, Su YN, Otoo A, Adu-Gyamfi EA, Feng Q, Wang YX, Wang MJ, Ding YB. Glycyrrhizin ameliorates impaired glucose metabolism and ovarian dysfunction in a polycystic ovary syndrome mouse model. Biol Reprod. 2023 Jul 11;109(1):83-96. doi: 10.1093/biolre/ioad048. PMID 37115805